CLINICAL TRIAL: NCT05815550
Title: Association Between Delirium and Use of Proton Pump Inhibitors: Analysis of the Global Pharmacovigilance Database
Brief Title: Delirium Related to Proton Pump Inhibitors Use
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2646
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2023-04

CONDITIONS: Proton Pump Inhibitor Adverse Reaction; Delirium; Hyponatremia
Keywords: Proton Pump Inhibitor; Delirium; Drug safety; Hyponatremia
MeSH Terms: conditions — Delirium; Hyponatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PPI users
  Interventions: Drug: PPI

INTERVENTIONS:
Drug: PPI — Use of PPI defined as PPI mentioned in the safety report

SUMMARY:
Delirium is a frequent and severe condition, especially in old adults. Its occurrence is due to a drug in 30% of cases. In 2009, the French national health authority (Haute Autorité de Santé) mentioned proton pump inhibitors (PPIs) among the drugs causing delirium. Most reports of delirium associated with PPI use in the literature are due to severe hyponatremia due to syndrome of inappropriate antidiuretic hormone secretion. However, a few case reports have described the occurrence of delirium PPI without hyponatremia related to PPI use. In 2016, a prospective observational study including 675 old adults found an association between PPI use and the occurrence of delirium.

Evidence linking delirium and PPI use is thus scarce. By using data from the pharmacovigilance database of the World Health Organization (WHO), the investigators aim to describe the characteristics of delirium reports in which PPI were suspected to be involved, and to evaluate the association between PPI use and delirium, and the impact of hyponatremia in this association by performing a disproportionality analysis.

ELIGIBILITY:
Inclusion Criteria:

* PPI use
* Delirium mentioned in the safety report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators describe the profile of patients who are reported in the WORLD HEALTH ORGANIZATION Vigibase pharmacovigilance database, as having experienced a delirium. In particular, the number of patients who use proton pomp inhibitors (PPIs), the number of patients who presented associated illnesses known to induce delirium, the number of patients who presented associated drug prescriptions known to induce delirium.
Sampling Method: Non-Probability Sample
Enrollment: 19081 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Delirium occuring when using PPI | 09/02/2022

SECONDARY OUTCOMES:
Association between PPI use and occurrence of delirium | 09/02/2022
  Association assessed by performing a disproportionality analysis with adjustment on confounders
Association between PPI use and occurrence of delirium and hyponatremia | 09/02/2022
  Association assessed by performing a disproportionality analysis with adjustment on confounders

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Decros A, Minoc EM, Lelong-Boulouard V, Chretien B, Meurant A, Alexandre J, Dolladille C, Villain C. Association between exposure to proton pump inhibitors and delirium: a descriptive and disproportionality analysis of VigiBase. BMJ Open. 2024 Oct 16;14(10):e081911. doi: 10.1136/bmjopen-2023-081911. PMID 39414279